CLINICAL TRIAL: NCT05366413
Title: Pilot Study of Early Referral to Interventional Pain Management for Patients With Advanced Malignancies
Brief Title: Early Interventional Treatment for Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Andrea Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-758
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cancer Pain
Keywords: Cancer Pain
MeSH Terms: conditions — Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Participants will receive early referral to an anesthesia-trained interventional pain management specialist evaluated for pain management strategies.
  Participants will complete surveys every 2 months and will have the option of tracking their pain at home using a secure smartphone application.
  Participants will be followed on the study for 4 months.
  Interventions: Other: Early Referral; Other: Pain Management Strategies

INTERVENTIONS:
Other: Early Referral — Directing a patient for a pain specialist consult earlier than standardly occurs.
Other: Pain Management Strategies — Specialized plan with procedures to ease pain

SUMMARY:
The purpose of the study is to evaluate how feasible and beneficial it is to refer patients with cancer pain to a doctor who specializes in pain management, including procedures to relieve pain, and whether this is helpful to patients with pain related to their cancer.

DETAILED DESCRIPTION:
This is a single arm pilot study evaluating a new system of referral and pain evaluation for patients with advanced solid tumors and moderate-to-severe pain who are not already on high-dose opioids to an anesthesia-trained interventional pain management specialist .

A variety of interventional treatments for pain have been proven effective for cancer patients. Often without early referral patients do not get evaluated for interventional procedures for their pain unless the pain is very severe, or they are admitted to the hospital. It is expect this intervention will work by providing effective pain treatments to patients sooner than they might normally be referred and will be evaluated by how many patients are candidates for interventional treatments for their pain, whether patients choose to receive these treatments, and whether patients find the pain specialist referral acceptable and helpful

The research study procedures include screening for eligibility, study interventions including evaluations and follow up visits, as well as surveys at the beginning, middle, and end of the study. Participants will be followed on the study for 4 months.

It is expected that about 30 people will take part in this research study.

Medtronic and is providing funding for this research study

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a metastatic, or locally advanced unresectable malignancy
* Anticipated prognosis of more than 6 months according to the primary oncologist
* Age greater than 21 years
* Persistent pain with an average pain rating of 4 or greater on an 11-point numeric rating scale (NRS) from 0-10 where 10 is considered the most severe.
* Pain has persisted for at least 2 weeks
* Pain is due to cancer or sequelae of cancer treatment

Exclusion Criteria:

* Primary pain syndrome is sensory peripheral neuropathy
* Patient is taking more than 200 morphine milligram equivalents (MMEs) per day on average, at the time of recruitment.
* Currently cared for by interventional pain management specialist
* Receipt of prior pain intervention (e.g. celiac neurolysis)
* Bleeding diathesis, uncontrollable infection, or other contra-indications to pain interventions
* History of opioid misuse disorder
* Inability to speak English
* Cognitive impairment or any other disorder that would impede study participation and survey completion
* If patients are unable to complete the baseline survey, they will no longer be considered eligible for the study; this will serve as an indication of barriers to participation that would make them unable to comply with study procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Pain Management Strategies: Participants will receive early referral to an anesthesia-trained interventional pain management specialist evaluated for pain management strategies.
  Participants will complete surveys every 2 months and will have the option of tracking their pain at home using a secure smartphone application.
  Participants will be followed on the study for 4 months.
  Early Referral: Directing a patient for a pain specialist consult earlier than standardly occurs.
  Pain Management Strategies: Specialized plan with procedures to ease pain
Period: Overall Study
Arm/Group | Pain Management Strategies
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pain Management Strategies
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59.5 [49.25 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Pain Consultation
Description: Feasibility will be measured by the percentage of patients that have an interventional pain consultation within 4 weeks, with a threshold for determining feasibility of at least 80% of participants.
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Arm: Participants will receive early referral to an anesthesia-trained interventional pain management specialist evaluated for pain management strategies.
  Participants will complete surveys every 2 months and will have the option of tracking their pain at home using a secure smartphone application.
  Participants will be followed on the study for 4 months.
  Early Referral: Directing a patient for a pain specialist consult earlier than standardly occurs.
  Pain Management Strategies: Specialized plan with procedures to ease pain
Arm/Group | Intervention Arm
Number analyzed (Participants) | 30
Participants | 29

2. Primary Outcome: Feasibility - Interventional Pain Procedure Rate
Description: Feasibility will be measured by the percentage of patients who ultimately receive at least one interventional pain procedure, with a threshold for determining feasibility of at least 50% of participants.
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 30
Participants | 18

3. Primary Outcome: Acceptability - Satisfaction Ratings
Description: Acceptability will be measured by the percentage of patients satisfied with their interventional pain management care, with a threshold of at least 80% of patients rating the quality of care received at the interventional pain management clinic at a 7 or above on a 0-10 scale (adapted from HCAHPS; 0 being the worst clinic possible, 10 being the best clinic possible). For participants with missing data at 4-months, we imputed their responses at 2-months.
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 18
Participants | 15

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pain Management Strategies
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT05366413/Prot_SAP_000.pdf